CLINICAL TRIAL: NCT02554695
Title: Effects of Age and Osteoclast Inhibition on Bone Formation
Brief Title: Osteoclast Inhibition and Bone Formation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sundeep Khosla, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 15-002313
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Bone Loss; Aging
Keywords: adrenergic
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Sodium Chloride; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): single subcutaneous injection of placebo (normal saline)
  Interventions: Drug: placebo
- Denosumab (Active Comparator): single subcutaneous injection of denosumab 60 mg
  Interventions: Drug: denosumab
- young normal premenopausal women (No Intervention): no intervention

INTERVENTIONS:
Drug: placebo — subcutaneous saline injection
  Other Names: saline
  Arms: placebo
Drug: denosumab — single subcutaneous injection of denosumab 60 mg
  Other Names: Prolia
  Arms: Denosumab

SUMMARY:
This protocol addresses: 1) How gene expression changes in bone cells are affected by aging? 2) Is aging associated with decreased signaling between bone cells? 3) How does treatment with the osteoporosis medication denosumab affect bone cell signaling?

DETAILED DESCRIPTION:
This protocol collectively addresses the following goals: 1) What are the changes in gene expression in osteoblasts and osteocytes that lead to impaired bone formation with aging; 2) Since recent work from the investigators' group has demonstrated that osteoclasts produce a number of growth factors and cytokines (coupling factors) that enhance osteoblast proliferation and/or differentiation, is aging associated with reduced osteoclast coupling factor production; and 3) If osteoclasts are markedly reduced using the FDA-approved medication for osteoporosis, denosumab, how does that effect the quantity of coupling factors in the bone microenvironment and the target genes of these coupling factors in osteoblasts?

ELIGIBILITY:
* Inclusion Criteria:

  * normal premenopausal women aged 25-40 years
  * normal postmenopausal women aged 60-80 years
  * at least 5 yrs since their last menses
  * follicle stimulating hormone (FSH) > 20 IU/L
* Exclusion Criteria:

  * Abnormality in any of the screening laboratory studies
  * Presence of significant liver or renal disease
  * Malignancy (including myeloma)
  * Malabsorption
  * Diabetes
  * Hypoparathyroidism
  * Hyperparathyroidism
  * Acromegaly
  * Cushing's syndrome
  * Hypopituitarism
  * Severe chronic obstructive pulmonary disease
  * Undergoing treatment with any medications that affect bone turnover, including the following:
* adrenocorticosteroids (> 3 months at any time or > 10 days within the previous yr)
* anticonvulsant therapy (within the previous year)
* pharmacological doses of thyroid hormone (causing decline of thyroid stimulating hormone below normal)
* calcium supplementation of > 1200 mg/d (within the preceding 3 months)
* bisphosphonates (within the past 3 yrs)
* denosumab
* estrogen (E) therapy within the past year
* treatment with a selective E receptor modulator within the past year
* teriparatide within the past yr

  * Clinical history of osteoporotic fracture (vertebral, hip, or distal forearm)
  * Recent (within the past 6 months) fracture
  * Serum 25-hydroxyvitamin D levels of < 20 ng/ml

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
Gene expression changes in bone cells | 3 months
  Ratio of selected genes as expressed between each of the 3 arms (i.e. relative runx2 gene expression levels in each arm).

SECONDARY OUTCOMES:
Osteoclast-osteoblast coupling factor changes | 3 months
  Ratio of selected genes as expressed between each of the 3 arms (i.e. relative runx2 gene expression levels in each arm).

CONTACTS AND LOCATIONS:
Overall Officials: Sundeep Khosla, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States